CLINICAL TRIAL: NCT02926846
Title: Randomized Trial on Intravenous Antibiotics With Adjunctive Lavage for Severe Peritoneal-dialysis Related Peritonitis
Brief Title: IV Antibiotics With Lavage for Severe PD Peritonitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alice Ho Miu Ling Nethersole Hospital (Other)
Responsible Party: Principal Investigator, Steve Siu-Man Wong, Associate Consultant, Alice Ho Miu Ling Nethersole Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013.201
Record Dates: First submitted 2016-10-01; First posted 2016-10-06 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Peritonitis; Kidney Failure
Keywords: Peritoneal dialysis; Lavage
MeSH Terms: conditions — Peritonitis; Renal Insufficiency | interventions — Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lavage arm (Experimental): Intravenous vancomycin & gentamicin with adjunctive lavage
  Interventions: Drug: Intravenous vancomycin & gentamicin with adjunctive lavage
- Standard treatment arm (Active Comparator): Intraperitoneal vancomycin & gentamicin
  Interventions: Drug: Intraperitoneal vancomycin & gentamicin

INTERVENTIONS:
Drug: Intravenous vancomycin & gentamicin with adjunctive lavage — Intravenous vancomycin and gentamicin are administered, together with adjunctive lavage performed by automated peritoneal dialysis machine over 48 to 72 hours.
  (choice of antibiotic is adjusted in accordance with the microbiology report when available)
  Arms: Lavage arm
Drug: Intraperitoneal vancomycin & gentamicin — Intraperitoneal vancomycin and gentamicin are administered, with the usual continuous ambulatory peritoneal dialysis schedule maintained.
  (choice of antibiotic is adjusted in accordance with the microbiology report when available)
  Arms: Standard treatment arm

SUMMARY:
This is a randomized controlled trial to evaluate whether a switch to intravenous antibiotics with adjunctive lavage can improve the outcome of severe peritoneal dialysis related peritonitis.

DETAILED DESCRIPTION:
The standard treatment of peritoneal dialysis (PD) related peritonitis is intraperitoneal (IP) antibiotics. In severe cases not responding to the IP antibiotics treatment, timely Tenckhoff catheter removal is needed. There is no known adjunctive measure that can improve the clinical outcome of the patients suffering from severe PD peritonitis.

Based on the past experience in the investigators' center, switching IP to intravenous route of antibiotics administration, together with adjunctive lavage was proposed to improve the clinical outcome of severe PD peritonitis, in particular a possible improved catheter salvage rate. This method will be evaluated in the present clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent PD patients with age >= 18 years old suffering from PD peritonitis
* PD effluent white cell count >1090/mm2 on peritonitis day 3
* Lack of clinical response
* Informed consent available

Exclusion Criteria:

* PD peritonitis in association with exit site or tunnel infection
* Relapsing peritonitis (i.e. peritonitis caused by same organism within 4 weeks after completion of antibiotics therapy)
* Fungal peritonitis
* Mycobacterial peritonitis (both tuberculosis and non-tuberculosis species)
* Clinical suspicion of surgical peritonitis
* Penicillin- or cephalosporin allergy, that cefazolin and ceftazidime could not be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Peritoneal dialysate effluent (PDE) white cell count and bacterial culture | PDE is monitored every 48 hours, until white cell count <100/mm3 and bacterial culture is negative; assessed up to 3 weeks
Number of participants requiring Tenckhoff catheter removal | Tenckhoff catheter removal is arranged when there is no clinical response after 5 days of treatment

SECONDARY OUTCOMES:
Number of participants developing relapsing peritonitis | All participants are observed for any peritonitis within 4 weeks of completion of antibiotics treatment
Number of participants requiring hospitalization | All participants are observed for any hospitalization within 12 weeks of completion of antibiotics treatment

CONTACTS AND LOCATIONS:
Overall Officials: Siu-Man Wong, MBChB, FRCPC, Principal Investigator — Alice Ho Miu Ling Nethersole Hospital
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided